CLINICAL TRIAL: NCT01556867
Title: Evaluation of Two Strategies for Umbilical Cord Care : Dry Cord Care Versus Antiseptic on the Incidence of Omphalitis in Healthy Term Newborn
Acronym: NEOCORD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/10/06-U
Record Dates: First submitted 2012-02-17; First posted 2012-03-16 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Omphalitis
Keywords: Umbilical cord care; dry cord care; antiseptic; Omphalitis; umbilical cord drop; hospitalized in maternity hospital
MeSH Terms: interventions — Desiccation

ARMS (2):
- dry cord care (Active Comparator)
  Interventions: Other: Cord care by simple debridement (soaping, rinsing and drying)
- antiseptic care (Active Comparator)
  Interventions: Other: Cord care with the use of antiseptics

INTERVENTIONS:
Other: Cord care by simple debridement (soaping, rinsing and drying) — For children born during an experimental period of cord care will be done with a simple debridement (soaping and then rinsing and drying carefully)
  Arms: dry cord care
Other: Cord care with the use of antiseptics — For children born during a control period, cord care will be done with an antiseptic whose choice is left to the discretion of the healthcare team.
  In this essay, it opted not to impose an antiseptic. Indeed, the objective of the trial is to compare the two strategies for management of care.
  Arms: antiseptic care

SUMMARY:
At birth, the umbilical cord is cut, separating physically and symbolically the mother of his child. Before cord drop, umbilical area is a possible way of bacterial infection. Thus, umbilical cord infections constitute a major cause of neonatal morbidity and mortality in developing countries. In industrialized countries, omphalitis cases have almost disappeared whatever cord care strategies. At this day, care practices appear extremely different between countries, based more on habits and convictions that on evidence-based medicine. The investigators propose to conduct a non inferiority multicenter clustered crossed randomized study. Observations sessions will be performed on two consecutive periods of 5 months: 4 months of recruitment and 1 month follow-up. Main objective is to demonstrate that dry cord care practice would not expose to a higher risk of omphalitis than antiseptic based care approach. The purpose of NEOCORD study is a simplification of cord care for paramedical teams and parents, but also a significant reduction of costs in a medico-economic approach.

ELIGIBILITY:
Inclusion Criteria:

* Newborn > 36 weeks of gestation.
* Asymptomatic newborn hospitalization.
* Information and consent of parental or legal authority.

Exclusion Criteria:

* Outborn.
* Family or social environment considered incompatible with dry cord care by investigator from a hygienic point of view (no fixed abode etc…).
* Hospitalization in neonatal intensive care unit.
* Transfer to another maternity hospital.
* Gestational age less than or equal to 36 weeks of gestation.
* Serious Congenital Pathology.
* Opposition of parents.

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8698 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The incidence of occurrence of omphalitis within 28 days post-birth in omphalitis incidence in healthy newborn | 13 months
  The primary endpoint will correspond to the incidence of omphalitis occurred within 28 days post-birth.
  The omphalitis is defined as the presence of erythema or serous or purulent in-cord tissue or umbilical perished. The stages are described to investigators about watching information in a search for suspected omphalitis.
  This can be confirmed retrospectively by an Awards Committee composed of a Dermatopédiatre, a pediatrician and a pediatric surgeon.

SECONDARY OUTCOMES:
Occurrence of neonatal infection defined as any situation requiring hospitalization and antibiotics in the first month of life | 13 months
  The analysis of the occurrence of neonatal infection will be conducted using the same strategy as that used for the primary outcome measure.
Date of the fall of the umbilical cord | 13 months
  The analysis of time to drop cord will also be conducted as part of a hierarchical model by considering a quantitative endpoint. If necessary, a transformation will be applied to the data before analysis.
Description of bacterial flora in umbilical waning of omphalitis | 13 months
  Regarding the bacterial flora, the analysis will be descriptive.
Parental satisfaction | 13 months
  Parental satisfaction, rated using a scale of 0 to 10, will be analyzed using a hierarchical model for quantitative data.
Occurrence of an infection or néonatlale maternal postpartum | 13 months
  Finally, concerning data on the health of mother and child (maternal infection, pertussis vaccination, sleeping habits, diet of the child), the analysis is purely descriptive.
State immunization against pertussis parental | 13 months
Sleeping patterns of children in the first months of life | 13 months
  Description of the sleeping patterns
Diet of the child at day 28. | 13 months
  Description of the infant feeding

CONTACTS AND LOCATIONS:
Overall Officials: Christèle GRAS-LE GUEN, PH, Principal Investigator — Nantes University Hospital; Christophe SAVAGNER, PH, Principal Investigator — University Hospital, Angers; Patrick PLADYS, PU-PH, Principal Investigator — Rennes University Hospital; Elie SALIBA, PU-PH, Principal Investigator — CHU de Tours; Gisèle GREMMO-FREGER, PH, Principal Investigator — CHU de Brest; Emmanuelle DESCOMBES-BARROSO, PH, Principal Investigator — Poitiers University Hospital
Locations (6):
- France (6):
  - Dr SAVAGNER Christophe, Angers
  - Dr GREMMO-FREGER Gisèle, Brest
  - Dr GRAS-LEGUEN, Nantes
  - Dr DESCOMBES-BARROSO Emmanuelle, Poitiers
  - Pr PLADYS Patrick, Rennes
  - Pr SALIBA Elie, Tours

REFERENCES:
- [Derived] Gras-Le Guen C, Caille A, Launay E, Boscher C, Godon N, Savagner C, Descombes E, Gremmo-Feger G, Pladys P, Saillant D, Legrand A, Caillon J, Barbarot S, Roze JC, Giraudeau B. Dry Care Versus Antiseptics for Umbilical Cord Care: A Cluster Randomized Trial. Pediatrics. 2017 Jan;139(1):e20161857. doi: 10.1542/peds.2016-1857. PMID 28008096